CLINICAL TRIAL: NCT02395237
Title: An Open-label, Randomized, Two-treatment Crossover Bioequivalence Study Comparing Two Batches of the Same Fixed Dose Combinations Amaryl® M IR 2/1000 (Glimepiride/Metformin Hydrochloride Immediate Release Combination Tablet) in Fed Conditions in Healthy Male and/or Female Subjects.
Brief Title: COMPOUND (INN): HOE490O - GLIMEPIRIDE / METFORMIN HCl (Amaryl® M)0 (Glimepiride/Metformin Hydrochloride Immediate Release Combination Tablet) in Fed Conditions in Healthy Male and/or Female Subjects.
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Pharmaceutical Research Unit, Jordan (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BEQ14393
Record Dates: First submitted 2015-03-17; First posted 2015-03-23 (Estimated); Last update posted 2020-09-18 (Actual); Status verified 2015-03

CONDITIONS: Healthy
Keywords: Fed Conditions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Amaryl® M IR 2/1000 (manufactured in India) (Experimental): Investigational products :Reference formulation Trade Name: Amaryl® M IR 2/1000 (manufactured in India) Dosage Form: Film coated tablet 1x1 Active Substance: Glimepiride/metformine HCl 2 mg/1000 mg Manufacturer: Goa, India
  Interventions: Drug: : Amaryl® M IR 2/1000
- Amaryl® M IR 2/1000 (manufactured in Turkey) (Experimental): Dosage form: Film coated tablet 1x1 Active substance : Glimepiride/metformine HCl 2 mg/1000 mg Manufacturer: Zentiva TR, Lüleburgaz
  Interventions: Drug: : Amaryl® M IR 2/1000

INTERVENTIONS:
Drug: : Amaryl® M IR 2/1000

SUMMARY:
The purpose of this study is to assess, after single oral administration under fed conditions, the bioequivalence between the two batches of the same glimepiride/metformin hydrochloride (HCl) 2 mg/1000 mg fixed dose combination (FDC) tablets (immediate release combination tablet Amaryl® M IR 2/1000) manufactured in India and in Turkey.

DETAILED DESCRIPTION:
An open-label, randomized, two-treatment crossover bioequivalence study comparing two batches of the same fixed dose combinations Amaryl® M IR 2/1000 (glimepiride/metformin hydrochloride immediate release combination tablet) in fed conditions in healthy male and/or female subjects.

Primary Objective To assess, after single oral administration under fed conditions, the bioequivalence between the two batches of the same glimepiride/metformin hydrochloride (HCl) 2 mg/1000 mg fixed dose combination (FDC) tablets (immediate release combination tablet Amaryl® M IR 2/1000) manufactured in India and in Turkey.

Secondary Objective(s) To assess the safety (including hypoglycemic events) of the two FDC (Amaryl® M IR 2/1000) tablets.

Up to 50 healthy subjects are to be enrolled to have 46 subjects available for the final pharmacokinetic evaluation.

Study treatment:

In each period A single dose of glimepiride/metformin HCl 2mg/1000 mg FDC (manufactured in India) Or single dose of glimepiride/metformin HCl 2mg/1000 mg FDC (manufactured in Turkey) will be administered after breakfast.

PRIMARY AND SECONDARY ENDPOINT(S)

Primary Endpoint:

Glimepiride and metformin: Cmax and AUClast

Secondary Endpoint(s):

Glimepiride and metformin: AUC0-inf, tlag, tmax and t1/2z Safety

DURATION OF STUDY (per patient) Screening : up to 15 days Treatments periods: 4 days each including treatment day Wash-out period: 4 to 7 days Follow-up: 4 to 7 days Total study duration: 37 days

ELIGIBILITY:
Inclusion Criteria:

- Demography

1. Male subjects and female subjects of non-childbearing potential (post- menopausal or sterilized) aged 18 to 50 years inclusive.
2. Body weight between 50.0 and 95.0 kg, inclusive, if male, and between 40.0 and 85.0 kg, inclusive, if female, body mass index between 18.0 and 30.0 kg/m2, inclusive.

   * Health status
3. Certified as healthy by a comprehensive clinical assessment (detailed medical history (hypo-, hypertension, allergy, other diseases, major surgery, micturition, defecation, sleep, illness within the last 3 weeks prior start of the trial, registration of life style and habits (consumption of alcohol, nicotine, coffee, tea, coke, special diet, drug abuse) and complete physical examination (general state and abnormal findings per system: endocrine/metabolic, allergies, drug sensitivities, head, neck, eyes, ears, nose, throat, cardiovascular, respiratory, gastrointestinal, hepatic/biliary, urogenital, musculoskeletal, Iymph nodes, skin, and neurological/psychiatric).
4. Normal vital signs after 10 minutes resting in supine position:

   * 90 mmHg < systolic blood pressure (SBP) <140 mmHg
   * 45 mmHg < diastolic blood pressure (DBP) <90 mmHg
   * 40 bpm < heart rate (HR) <100 bpm
5. Normal standard 12-lead electrocardiogram (ECG) after 10 minutes resting in supine position in the following ranges; 120 ms<PR<220 ms, QRS<120 ms, QTc≤430 ms if male, ≤450 ms if female and normal ECG tracing unless the Investigator considers an ECG tracing abnormality to be not clinically relevant.
6. Laboratory parameters within the normal range (or defined screening threshold for the Investigator site), unless the Investigator considers an abnormality to be clinically irrelevant for healthy subjects; however blood/serum examination creatinine, alkaline phosphatase, hepatic enzymes (aspartate aminotransferase, alanine aminotransferase), and total bilirubin (unless the subject has documented Gilbert syndrome) should not exceed the upper laboratory norm. For female of non-childbearing potential, sterilized at least 3 months earlier or postmenopausal i.e. artificial or natural menopause for more than 2 years with plasma FSH level > 30 UI/L.

Regulations I 07. Having given written informed consent prior to undertaking any study-related procedure.

I 08. Covered by a health insurance system where applicable, and/or in compliance with the recommendations of the national laws in force relating to biomedical research.

I 09. Not under any administrative or legal supervision.

Exclusion Criteria:

* Medical history and clinical status E 01. Any history or presence of clinically relevant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic, hematological, neurological, osteomuscular, articular, psychiatric, systemic, ocular, gynecologic (if female), or infectious disease, or signs of acute illness.

E 02. Frequent headaches and/or migraine, recurrent nausea and/or vomiting (more than twice a month).

E 03. Blood donation, any volume, within 3 months before inclusion. E 04. Symptomatic hypotension, irrespective of the decrease in blood pressure. E 05. Presence or history of drug hypersensitivity, or allergic disease diagnosed and treated by a physician.

E 06. Major surgery of the gastrointestinal tract except for appendectomy. E 07. History or presence of drug or alcohol abuse (alcohol consumption more than 40 g per day).

E 08. Smoking more than 5 cigarettes or equivalent per day, unable to stop smoking during the study.

E 09. Excessive consumption of beverages containing xanthine bases (Pepsi/cola, tea, coffee) more than 4 cups or glasses per day) E 10. If female, pregnancy (defined as positive β-HCG test), breast-feeding. Interfering substance E 11. Medication with drugs known to alter organs or systems such as barbiturates, phenothiazines, cimetidine, omeprazole etc. within the last 2 months.

E 12. Any medication (including St John's Wort) within 14 days before inclusion or within 5 times the elimination half-life or pharmacodynamic half-life of the medication, any vaccination within the last 28 days and any biologics (antibody or its derivatives) given within 4 months before inclusion.

General conditions E 13. Any subject who, in the judgment of the Investigator, is likely to be noncompliant during the study, or unable to cooperate because of a language problem or poor mental development.

E 14. Any subject in the exclusion period of a previous study according to applicable regulations.

E 15. Any subject who cannot be contacted in case of emergency. E 16. Any subject who is the Investigator or any subinvestigator, research assistant, pharmacist, study coordinator, or other staff thereof, directly involved in conducting the study.

Biological status E 17. Positive result on any of the following tests: hepatitis B surface (HBs Ag) antigen, anti-hepatitis C virus (anti-HCV) antibodies, anti-human immunodeficiency virus 1 and 2 antibodies (anti-HIV1 and anti HIV2 Ab).

E 18. Positive result on urine drug screen (amphetamines/methamphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, opiates).

E 19. Positive alcohol test. Specific to the study E 20. Any contra-indications to glimepiride, according to the applicable labeling.

E 21. Any contra-indications to metformin, according to the applicable labeling.

E 22. Use of any CYP2C9 inhibitors and/or CYP2C9 inducers within 7 days before inclusion.

E 23. Vegetarian diet E 24. Participation in another clinical trial at same time or within the preceding 3 months (calculated from the date of the final examination of the previous study),except for previous BE trials in which case 80 days are sufficient.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Cmax | 0-72
AUC0-t | 0-72

SECONDARY OUTCOMES:
AUC0-inf | 0-72

CONTACTS AND LOCATIONS:
Locations (1):
- Arab Pharmaceutical industry Consulting/ Pharmaceutical Research Unit, Amman, Jordan